CLINICAL TRIAL: NCT06063291
Title: A Randomized, Double-blinded, Placebo-controlled, Single Ascending Dose Phase 1 Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetics After a Single Oral Administration of ID110521156 in Healthy Subjects
Brief Title: Single Ascending Oral Dose Phase 1 Study of ID110521156 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Collaborators: YUNOVIA CO.,LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: ID110521156-T2DM-101
Record Dates: First submitted 2023-09-13; First posted 2023-10-02 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1 will consist of 8 healthy subjects who will be randomised to receive a single oral dose of ID110521156 of placebo.
  Interventions: Drug: ID110521156; Drug: Placebo of ID110521156
- Cohort 2 (Experimental): Cohort 2 will consist of 8 healthy subjects who will be randomised to receive a single oral dose of ID110521156 of placebo.
  Interventions: Drug: ID110521156; Drug: Placebo of ID110521156
- Cohort 3 (Experimental): Cohort 3 will consist of 8 healthy subjects who will be randomised to receive a single oral dose of ID110521156 of placebo.
  Interventions: Drug: ID110521156; Drug: Placebo of ID110521156
- Cohort 4 (Experimental): Cohort 4 will consist of 12 healthy subjects who will receive a single oral dose of ID110521156 at fed state and fasted state each.
  Interventions: Drug: ID110521156

INTERVENTIONS:
Drug: ID110521156 — subjects will receive a single oral dose of IMP. In the morning (all procedures must be performed at the similar clock time) on Day 1
Drug: Placebo of ID110521156 — subjects will receive a single oral dose of IMP. In the morning (all procedures must be performed at the similar clock time) on Day 1
  Arms: Cohort 1; Cohort 2; Cohort 3

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of single oral doses of ID110521156 in healthy adult subjects. This is the first clinical study of ID110521156.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 19 to 50 years at the time of Screening.
* Body mass index (BMI) within 18.5 to 29.9 kg/m2; and a total body weight ≥ 40 kg, ≤ 90 kg
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* For female subjects, not pregnant or lactation women, or naturally menopausal (spontaneous amenorrhea for at least 12 months) or surgically infertility (bilateral tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy etc).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal(including pancreatitis), cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing.
* Treatment with an investigational drug (including a bioequivalence study) within 6 months prior to the scheduled date of administration of the investigational product.
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 3 months after the last dose.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
AEs/serious AEs (SAEs) | Throughout study duration, up to 9 days
  Incidence and severity of ad adverse event
Percentage of subjects with clinically significant change from baseline in vital signs, ECG, safety laboratory test results | Throughout study duration, up to 9 days

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Area under the plasma drug concentration-time curve from 0 to last, (AUClast) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Area under the plasma drug concentration-time curve from 0 to infinity (AUCinf) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
The time of peak concentration,(Tmax) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Terminal half-life (T1/2) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Apparent clearance (CL/F) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Apparent volume of distribution after extravascular administration (Vd/F) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Amount excreted in urine (Ae) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Renal Clearance (CLr) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156
Fraction excreted unchanged of an administered dose (fe) | Throughout study duration, up to 9 days
  Both plasma and urine PK of ID110521156 will be assessed after single dose administration of ID110521156

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided